CLINICAL TRIAL: NCT05556356
Title: Effect of Perioperative Acetaminophen Dosing on Patients Undergoing Surgical Treatment of Basilar Thumb Arthritis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Physician decision
Sponsor: Indiana Hand to Shoulder Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IU15386
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Carpometacarpal Osteoarthritis
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants unblinded following final data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group (Placebo Comparator): Preoperative multivitamin and postoperative standardized pain management regimen
  Interventions: Other: Placebo: Multivitamin
- Test Group (Experimental): : Preoperative acetaminophen and postoperative standardized pain management regimen
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — pre-operative acetaminophen (1000mg)
  Other Names: Tylenol
  Arms: Test Group
Other: Placebo: Multivitamin — pre-operative Multivitamin
  Arms: Control Group

SUMMARY:
Basilar thumb arthritis is a common problem that affects 7% of men and 15% of women. It is regarded as one of the more painful procedures commonly performed by hand surgeons. Opioid overuse and diversion are significant problems in the country that contribute to opioid addiction as well as deaths from opioid overdose. Prior studies have examined the effect of different nerve block compositions on perioperative and postoperative analgesia, but none have looked at perioperative loading analgesia. We will attempt to address this problem by exploring alternative analgesia regimens to decrease opioid prescribing after 1st carpometacarpal (CMC) joint arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or older)
* Patients presenting with symptomatic 1st CMC arthritis with or without scaphotrapeziotrapezoid arthritis
* Eaton Classification stage II, III, or IV OA of the first CMC joint based on xrays
* Patients who plan to undergo a ligament reconstruction and tendon interposition (LRTI) or thumb suspensionplasty procedure within 6 months of enrolling to study
* Bilateral thumbs included

Exclusion Criteria:

* <18 years age
* Prior surgical history of ipsilateral 1st CMC arthroplasty or procedures involving thumb CMC joints
* Prior ipsilateral tendon rupture or ipsilateral peripheral nerve palsy
* History of opioid dependency or current chronic opioid use
* Contraindication to acetaminophen use
* Contraindication to NSAID use
* Contraindication or known allergy to peripheral nerve blockade, including coagulopathy
* Contraindication to supraclavicular block due to anatomic variability or inability to tolerate phrenic nerve blockade.
* Contraindication to multivitamin use
* Liver dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 2 weeks
  Patients report pain on a scale of 0 (no pain) to 100 (worst possible pain)
Number of Narcotic Pills Used | 2 weeks
  Number of Narcotic Pills Used

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana Hand to Shoulder Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No